CLINICAL TRIAL: NCT03686306
Title: VIRTUOSE : Efficiency of Sildenafil on the Absolute Claudication Distance of Peripheral Arterial Disease Patients With Intermittent Claudication. A Phase III, National, Multicentre, Prospective, Randomised, Double-blind, Placebo-Controlled Trial.
Brief Title: VIRTUOSE : Efficiency of Sildenafil on the Absolute Claudication Distance of Peripheral Arterial Disease Patients With Intermittent Claudication.
Acronym: VIRTUOSE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIRTUOSE; 2020-000231-42 (EudraCT Number); 20 07 41 (Other: CPP); MEDAECNAT-2020-07- 00008 (Other: ANSM)
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Experimental design A Phase III, National, Multicentre, Prospective, Randomised, Double Blind, placebo-controlled clinical trial with two parallel groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The preparation of the 'blinded' treatments will be undertaken by the PPRIGO hospital pharmacist's consortium (Production Pharmaceutique pour la Recherche Institutionnelle du Grand Ouest) under recommended standardised conditions. PPRIGO will provide numbered and labelled boxes each containing 32 capsules of the study drug (sildenafil or placebo according to the randomisation order). All boxes will be identically labelled, with the study number being the only differentiating feature between different drug packs.
  The un-blinding will be centralised with eCRF software in agreement with the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Sildenafil citrate 140 mg/day (single morning oral dose of 140 mg) for a total duration of 24 weeks.
  Interventions: Drug: Sildenafil
- Control group (Placebo Comparator): Placebo (single morning oral dose) for a total duration of 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil citrate 140 mg/day (single morning oral dose of 140 mg) for a total duration of 24 weeks. + advice to walk for a total duration of 6 months.
  Treatment will be proposed in addition to optimal treatment (Antiplatelet + Lipid Lowering Drugs + AT2 antagonists / ACE Inhibitors; unless contra-indicated) + advice to walk.
  Arms: Experimental group
Drug: Placebo — Placebo (single morning oral dose) + advice to walk for a total duration of 24 weeks.
  Treatment will be proposed in addition to optimal treatment (Antiplatelet / Direct Oral Anticoagulant + Lipid Lowering Drugs + AT2 antagonists / ACE Inhibitors; unless contra-indicated) + advice to walk.
  Arms: Control group

SUMMARY:
Peripheral Arterial Disease (PAD) is a highly debilitating disease that affects 202 million people around the world and about 7 million people in France. Morbi-mortality from cardiovascular events is increased in this population. Intermittent claudication is defined as a discomfort and/or pain in the legs during walking. It is the most common clinical feature of PAD.

In claudication, primary therapeutic approach is medical treatment and advice to walk. Revascularization is only proposed when medical treatment and advice to walk for at least 3 to 6 months have failed to improve symptoms and walking ability.

Optimal medical treatment includes Antiplatelet, Lipid Lowering Drugs, AT2 antagonists / ACE Inhibitors and advice to walk.

To date, no other drug has provided consistent evidence for functional improvement in claudication, except for Cilostazol, a type-3 phospho-diesterase inhibitor (PDEi). This compound has been scarcely used in France due to cost and frequent side effect (Headache, Flush, Diarrhea, etc.) and was withdrawn as a therapy in 2010.

Sildenafil, a type 5 PDEi, is well tolerated, largely used in impotence and has interesting clinical delay and duration of action in the concept of a potential use in claudication. Preliminary data from the literature and unpublished case reports, suggest that this drug could efficiently improve symptoms and walking capacity in patients with stage 2 claudication.

DETAILED DESCRIPTION:
Experimental design A Phase III, National, Multicentre, Prospective, Randomised, Double Blind, placebo-controlled clinical trial with two parallel groups.

Eligible patients will be randomised in two groups:

* Experimental group Sildenafil citrate 140 mg/day (single morning oral dose of 140 mg) for a total duration of 24 weeks.
* Control group Placebo (single morning oral dose) for a total duration of 24 weeks.

Treatment will be proposed in addition to optimal treatment (Antiplatelet / Direct Oral Anticoagulant + Lipid Lowering Drugs + AT2 antagonists / ACE Inhibitors; unless contra-indicated) + advice to walk.

The experimental drug will be delivered for a 4 weeks treatment period. Phone contact will be carried out at 7 and 14 days focusing on tolerance, compliance and eventual side effects.

First follow up visit at week 4 will focus on tolerance, compliance and side effects. If no major side effect is found, the study drug will be delivered for an additional 8 weeks.

Phone contact will be carried out at 8 weeks focusing on tolerance, compliance and eventual side effects.

Patients will be evaluated at week 12 (second follow-up visit) for persistent or non-persistent indication for revascularization and considered for revascularization if needed. In parallel, attention will be given to tolerance, compliance and eventual side effects. If no major side effect is found, the study drug will be delivered for an additional 12 weeks period.

Phone contact will be carried out at weeks 16 and 20 focusing on tolerance, compliance and eventual side effects.

Third and fourth follow-up visits are scheduled at week 24 (end of treatment) and week 48 (24 weeks after the end of experimental drugs).

Perspectives

* Improving quality of life of patients suffering a chronic debilitating disease is a major issue not only in vascular medicine.
* It is expected that the treatment may help patients change from a vicious circle (Pain > inactivity > disease progression > pain > increased morbi-mortality) to a virtuous circle (no Pain > improved ability for activity > collateral vessel development > slowing of disease progression > decreased morbi-mortality )
* We expect that half of the patients that fulfil inclusion criteria will be sufficiently improved not to require surgery anymore even 24 weeks after the end of the drug as a result of this virtuous circle.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old;
2. with peripheral artery disease (ABI ≤ 0.90 or TBI ≤ 0.70 or post-exercise ABI decrease of 18.5% from rest or ABI Exercise TcPO2 with DROPmin ≤ - 15 mmHg) reporting stable limiting claudication despite optimal medical treatment (Antiplatelet / Direct Oral Anticoagulant + Lipid Lowering Drugs + AT2 antagonists / ACE Inhibitors; unless contra-indication) and advice to walk for at least 4 weeks;
3. with a walking capacity lower or equal to 500 meters on treadmill;
4. affiliation to a social security agency
5. Patient who has understood the protocol and signed the consent form to participate.

Exclusion Criteria:

1. Revascularization already decided and scheduled;
2. Critical limb ischemia;
3. Life threatening disease;
4. Contraindication related to Sildenafil:

   * Patients treated with nitrates or drugs interfering with the action of sildenafil
   * Ongoing treatment by Ritonavir or alpha-blockers
   * Hypersensitivity to sildenafil or any of the excipients (lactose monohydrate)
   * Recent history of myocardial infarction or stroke < 3 months
   * Severe cardiovascular disorders such as unstable angina, severe cardiac failure and cardiomyopathy
   * Hypotension (Blood pressure < 90/50 mmHg)
   * Severe renal or hepatic failure
   * Amblyopia
   * Loss of vision in one eye because of Non-arterial ischemic Ophtalmic Neuropathy (NAION)
   * Known hereditary degenerative retinal disorders such as retinitis pigmentosa
   * Leukemia, Drepanocytosis, Multiple Myeloma
5. Pregnancy or breastfeeding;
6. Subjects under reinforced protection, deprived of liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social care establishment for purposes other than research;
7. Being in an exclusion period for another clinical study or in an ongoing interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Absolute claudication distance | Baseline and week 24
  Absolute change of the absolute claudication distance (ACD) from baseline to week 24

SECONDARY OUTCOMES:
Surgical re-vascularisation | baseline and weeks 24 and 48
  Rate of patients with surgical re-vascularisation at weeks 24 and 48
ACD | Baseline and week 48
  Absolute change of the ACD from baseline to week 48
Event free survival (EFS) | Through the study completion, an average of 1 year
  An "EVENT" is defined as either (1) major adverse cardiovascular events (MACE; including vascular deaths, non-fatal myocardial infarction and non-fatal stroke), (2) leg amputations, (3) Non Cardiovascular death.
  Event-free survival is defined as the time from inclusion to the first documented event. If no event is observed, event-free survival is defined as the delay of follow-up.
36-Item Short Form Health Survey (SF36) | Baseline and weeks 12, 24 and 48
  Quality of life : SF36 questionnaire at baseline and weeks 12, 24 and 48
Peripheral Artery Questionnaire | Baseline and weeks 12, 24 and 48
  Peripheral Artery Questionnaire at baseline and weeks 12, 24 and 48
Oxymetry | Baseline and weeks 12, 24 and 48
  Change in exercise oxymetry results between baseline and weeks 12, 24 and 48
Endothelial function by Laser Speckle | Baseline and weeks 12, 24 and 48
  Change in endothelial function at weeks 12, 24 and 48
Pulmonary function | Baseline and week 24
  Pulmonary function and diffusion capacity of the lungs for carbon monoxide (DLCO) at week 24 from baseline
Respect of prescribed dose | Through the study completion, an average of 1 year
  Compliance with the treatment
Tolerance | Through the study completion, an average of 1 year
  Tolerance and side effects
Arterial stifness | Baseline and weeks 12, 24 and 48
  Changes in arterial stiffness (Pulse Wave Velocity) with pOpmetre® between baseline and weeks 12, 24 and 48
Central Blood Pressure | Baseline and weeks 12, 24 and 48
  Changes in Central Blood Pressure with pOpmetre® between baseline and weeks 12, 24 and 48
Arterial compliance | Baseline and weeks 12, 24 and 48
  Changes in arterial compliance with Finometer® between baseline and weeks 12, 24 and 48
Vascular resistance | Baseline and weeks 12, 24 and 48
  Changes in vascular resistance with Finometer® between baseline and weeks 12, 24 and 48
Metabolomics signature | Baseline and week 24
  Change in metabolomics signature between baseline and week 24

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Guillaume MAHE, Rennes, Brittany Region
  - Amiens University Hospital, Amiens
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Cholet Hospital, Cholet
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Grenoble University Hospital, Grenoble
  - Mulhouse Hospital, Mulhouse
  - Nîmes University Hospital, Nîmes
  - AP-HP - Hôpital Européen Georges Pompidou, Paris
  - Hospital Paris Saint-Joseph and Hospital Marie Lannelongue, Paris

IPD SHARING:
Plan to Share IPD: No